CLINICAL TRIAL: NCT03966300
Title: Playing CARDs to Improve the Vaccination Experience at School: a Cluster Randomized Controlled Trial
Brief Title: Improving the School Vaccination Experience: What CARDs Are You Going to Play?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to inability to: 1) vaccinate at school, 2) control and track vaccinations, 3) continue the intervention as proposed. Data collected during fall 2019 clinics are being transferred to researchers and verified.
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37598
Record Dates: First submitted 2019-05-25; First posted 2019-05-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Vaccine Adverse Reaction; Vaccination; Complications; Fear
Keywords: school vaccinations; pain management; vaccination hesitancy; knowledge translation
MeSH Terms: conditions — Agnosia; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial; schools will be randomized to CARD or usual care and all students attending the schools will receive the allocated treatment
Who Masked: Participant
Masking Description: Students will not be aware of whether they are in the intervention or control group. Care providers who are trained in the intervention are aware of the group allocation. They will not communicate with care providers not trained in the intervention. Care providers that are trained in the intervention will not deliver care to participants in the control group and care providers that are not trained will not deliver care to participants in the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARD (multi-faceted knowledge translation intervention) (Experimental): CARD will be integrated into the school vaccination program. This includes pre-vaccination day preparation (e.g., planning of clinic spaces, student and school staff education about CARD) and vaccination day activities (e.g., clinic set-up, processes for triaging students, implementing pain/fear/fainting mitigation interventions from CARD during vaccination)
  Interventions: Other: Multi-faceted knowledge translation intervention
- Control (standard/usual care) (No Intervention): There are no specific procedures being undertaken to plan or execute clinics. Usual practices will be instituted (i.e., no education specific to CARD, nor clinic set-up or execution to incorporate interventions for pain, fear or fainting)

INTERVENTIONS:
Other: Multi-faceted knowledge translation intervention — The intervention consists of education of relevant stakeholders of best practices and integration of best practices into the vaccination delivery program
  Other Names: CARD
  Arms: CARD (multi-faceted knowledge translation intervention)

SUMMARY:
Vaccination hesitancy is identified as a threat to global health by the World Health Organization (WHO). For adolescents undergoing vaccination at school, prior studies demonstrate that concerns about pain and/or fear of needles contribute to negative experiences with vaccination and non-compliance with vaccination. The investigators developed an intervention that addresses vaccination hesitancy. In this study, investigators will evaluate the effectiveness of this intervention in a randomized controlled trial.

DETAILED DESCRIPTION:
Vaccination hesitancy is identified by the World Health Organization (WHO) as one of ten threats to global health. The WHO's 3C model of vaccination hesitancy identifies 3 domains of vaccine hesitancy: 1) Confidence (trust in health care providers), 2) Complacency (perceived importance of vaccine-preventable disease) and 3) Convenience (improving clinic processes). The investigators developed a multifaceted knowledge translation intervention that addresses vaccination hesitancy in school-based vaccinations. The intervention is called The CARD(TM) System (C-Comfort, A-Ask, R-Relax, D-Distract). CARD is a framework for delivering vaccinations that is student-centred and promotes coping. CARD integrates evidence-based interventions related to planning and execution of school vaccination clinics to directly tackle all 3 domains of vaccination hesitancy. It tackles Confidence by improving pain/fear management (it teaches students and public health staff how to reduce student symptoms which improves the vaccination experience and improves student trust in health care providers). It tackles Complacency by educating students about what vaccines are, why they are needed, community immunity, as well as the specific diseases they are being protected against. It tackles Convenience by improving school-based clinic processes by integrating student preferences (e.g., privacy, having a support person present).

In this randomized controlled trial, the investigators will evaluate the impact of CARD (vs. usual care) on student important outcomes and process outcomes.

ELIGIBILITY:
Inclusion Criteria:

* grade 7 students eligible for vaccination at school
* public health staff working in the school vaccination program

Exclusion Criteria:

* unable to understand and read English

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1919 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Student fear | within 5 minutes after vaccination
  student self-reported fear during vaccination, rated on a 0-10 scale

SECONDARY OUTCOMES:
Student pain | within 5 minutes after vaccination
  student self-reported pain during vaccination, rated on a 0-10 scale
Student dizziness | within 5 minutes of vaccination
  student self-reported dizziness during vaccination, rated on a 0-10 scale
Student fainting | within 1 hour after vaccination
  student fainting during vaccination, yes/no, as assessed by immunizer
Student post-immunization stress-related responses | within 1 hour after vaccination
  student post-immunization stress-related responses, yes/no, as assessed by immunizer using the WHO immunization Stress Responses Criteria
Utilization of coping strategies | within 5 minutes after vaccination
  use of individual coping strategies during vaccination (distraction, topical anesthetic, privacy, support person, deep breathing, muscle tension), yes/no, as assessed by immunizer using Documentation Checklist
Uptake of vaccination | by end of school year
  proportion of students vaccinated (overall and for each vaccine)
Implementation success of CARD | within 3 months of vaccination clinics
  perceptions of implementation success of CARD program delivery as reported by CARD implementers (primary targets) using the CARD Global Impression Checklist, individual questions (5-point likert scale, higher number represents better outcome). This information will be supplemented with information from focus groups with implementers and study notes
Compliance with CARD | within 3 months of vaccination clinics
  percent compliance with CARD implementation as assessed by implementers using a CARD compliance checklist. This information will be supplemented with information from focus groups with implementers and study notes
Knowledge of effective coping strategies | within 3 months after vaccination clinics
  knowledge of effective coping strategies, as assessed using a 10-point investigator-developed knowledge test, administered to implementers
Perceptions about pain and fear | within 3 months of vaccination clinics
  perceptions about pain and fear, as assessed using a 5-point likert scale (higher number represents better outcome) for implementers
Perceptions about vaccination program | within 3 months of vaccination clinics
  perceptions about vaccination program, as assessed using the Vaccination Program Global Impresssion Checklist, individual questions (5-point likert scale, higher number represents better outcome) for implementers
Willingness to be vaccinated | within 5 minutes after vaccination
  student self-reported willingness to be vaccinated, as assessed using a 5-point likert scale (higher number represents better outcome)
Satisfaction with CARD | within 5 minutes after vaccination
  student self-reported satisfaction with CARD, as assessed using Student Feedback Survey, individual questions (5-point likert scale, higher number indicates better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Wellington Dufferin Guelph Public Health, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Taddio A, Gudzak V, Jantzi M, Logeman C, Bucci LM, MacDonald NE, Moineddin R. Impact of the CARD (Comfort Ask Relax Distract) system on school-based vaccinations: A cluster randomized trial. Vaccine. 2022 Apr 26;40(19):2802-2809. doi: 10.1016/j.vaccine.2022.02.069. Epub 2022 Mar 29. PMID 35365344